CLINICAL TRIAL: NCT02354157
Title: Field Observation of Adverse Nutritional Effect of Parental Use of Food as a Reinforcer for Non-food Related Behavior
Brief Title: The Nutritional Effect of Parental Use of Food as a Reward
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Laurette Dube, Professor, McGill University
Other Study IDs: SSHRC-Insight: 435-2014-1964
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Children's Nutrition Intake
Keywords: children dietary pattern; control rules; instrumental learning; food reinforcement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Control rules are common parental practices that use food as reward to encourage children to conduct parents' preferred behaviors. This field observational study aims to examine whether control rules are associated with children's increased fat, carbohydrate and total energy intake in everyday eating, and whether this effect is moderated by individual differences in sensitivity to reward, and by gender differences.

DETAILED DESCRIPTION:
Control rules are parental practices that use food as an instrumental reinforcer to encourage children to behave in a normative manner in non-food domains. Since food high in fat or sugar is usually chosen as a reinforcer for control rules, these rules may lead to children's increased preference and every day intake of food high in sugar/fat. Research propositions were examined in 207 six to twelve-year-old children (97 boys and 110 girls). Their parents reported the children's everyday dietary intake through a food frequency questionnaire, and provided information regarding the children's sensitivity to rewards as well as an indication of how frequently they enforce family control rules.

ELIGIBILITY:
Inclusion Criteria:

* participants have 6-12 years old children

Exclusion Criteria:

* N.A.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The parents or guardians of 207 children (97 boys and 110 girls) aged from 6 to 12 (M=8.98, SD=1.67) completed the study. Participants were recruited from metropolitan Montreal, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Food Frequency Questionnaire | last month recall
  A web-based Food Frequency Questionnaire was used to aske participants' parents to recall their children's food intake over the last month based on a list of 136 individual food items or food clusters, which covered eight categories of food and beverages. For each individual food item or cluster, participants were asked to indicate how frequently their children consumed that food and the typical portion size.